CLINICAL TRIAL: NCT04562389
Title: A Phase 1/3 Study to Evaluate Efficacy and Safety of Selinexor, a Selective Inhibitor of Nuclear Export, in Combination With Ruxolitinib in Treatment-naïve Patients With Myelofibrosis
Brief Title: Study of Selinexor in Combination With Ruxolitinib in Myelofibrosis
Acronym: SENTRY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XPORT-MF-034; 2020-003883-19 (EudraCT Number); 2023-506139-13-00 (EU CTIS Number)
Record Dates: First submitted 2020-09-14; First posted 2020-09-24 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Selinexor; Ruxolitinib; Janus kinase 2; Myeloproliferative neoplasms
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders | interventions — selinexor; ruxolitinib

STUDY DESIGN:
Intervention Model Description: Phase 1, open-label, selinexor dose escalation and expansion part (enrollment completed). Phase 3, randomized, double-blind, placebo-controlled part.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 1a: Cohort 1: Selinexor 40 mg + Ruxolitinib BID (Experimental): Participants with MF will receive a dose of 40 milligrams (mg) selinexor oral tablets once weekly (QW) on Days 1, 8, 15, and 22 of each 28-day cycle in combination with 15 or 20 mg ruxolitinib twice a day (BID) based on the participants baseline platelet count.
  Interventions: Drug: Selinexor; Drug: Ruxolitinib
- Phase 1a: Cohort 2: Selinexor 60 mg + Ruxolitinib BID (Experimental): Participants with MF will receive a dose of 60 mg selinexor oral tablets QW on Days 1, 8, 15, and 22 of each 28-day cycle in combination with 15 or 20 mg ruxolitinib BID based on the participants baseline platelet count.
  Interventions: Drug: Selinexor; Drug: Ruxolitinib
- Phase 1b: Selinexor and Ruxolitinib BID (Experimental): Participants with MF will receive a dose of 40 or 60 mg selinexor oral tablets QW on Days 1, 8, 15, and 22 of each 28-day cycle in combination with 15 or 20 mg ruxolitinib BID based on the participants baseline platelet count.
  Interventions: Drug: Selinexor; Drug: Ruxolitinib
- Phase 3: Selinexor 60 mg + Ruxolitinib BID (Experimental): Participants with MF will receive a fixed starting dose of 60 mg selinexor (RD) oral tablets QW on Days 1, 8, 15, and 22 of each 28-day cycle in combination with a starting dose of 15 or 20 mg ruxolitinib BID based on the participants baseline platelet count.
  Interventions: Drug: Selinexor; Drug: Ruxolitinib
- Phase 3: Placebo + Ruxolitinib BID (Active Comparator): Participants with MF will receive a matching placebo of selinexor oral tablets QW on Days 1, 8, 15, and 22 of each 28-day cycle in combination with a starting dose of 15 or 20 mg ruxolitinib BID based on the participants baseline platelet count.
  Interventions: Other: Placebo; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Selinexor — Participants will receive a dose of 40 or 60 mg selinexor oral tablets QW.
  Other Names: KPT-330
  Arms: Phase 1a: Cohort 1: Selinexor 40 mg + Ruxolitinib BID; Phase 1a: Cohort 2: Selinexor 60 mg + Ruxolitinib BID; Phase 1b: Selinexor and Ruxolitinib BID
Drug: Selinexor — Participants will receive a dose of 60 mg selinexor oral tablets QW.
  Other Names: KPT-330
  Arms: Phase 3: Selinexor 60 mg + Ruxolitinib BID
Other: Placebo — Participants will receive a matching placebo of selinexor oral tablets QW
  Arms: Phase 3: Placebo + Ruxolitinib BID
Drug: Ruxolitinib — Participants will receive a dose of 15 or 20 mg ruxolitinib oral tablets BID.

SUMMARY:
This is a global, multicenter, 2-part study to evaluate the efficacy and safety of selinexor plus ruxolitinib in JAK inhibitor (JAKi) treatment-naïve myelofibrosis (MF) participants. The study will be conducted in two phases: Phase 1 (open-label) and Phase 3 (double-blind). Phase 1 (enrollment completed) was an open-label evaluation of the safety and recommended Phase 2 dose (RP2D) of selinexor in combination with ruxolitinib and included a dose escalation using a standard 3+3 design (Phase 1a) and a dose expansion part (Phase 1b). Phase 3 (ongoing), double-blind, placebo-controlled part of the study comparing the efficacy and safety of combination therapy of selinexor + ruxolitinib with combination of placebo + ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* A diagnosis of primary MF or post-essential thrombocythemia (ET) or postpolycythemia- vera (PV) MF.
* Active symptoms of MF as determined by presence of at least 2 symptoms using the Myelofibrosis Symptom Assessment Form (MFSAF) V4.0.
* Participants with international prognostic scoring system (DIPSS) risk category of intermediate-1, or intermediate-2, or high-risk.
* Measurable splenomegaly during the screening period as demonstrated by spleen volume of greater than or equal to (>=) 450 cubic centimeter (cm^3) .
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to (<=) 2.

Exclusion Criteria:

* More than 10% blasts in peripheral blood or bone marrow (accelerated or blast phase).
* Previous treatment with JAK inhibitors for MF.
* Previous treatment with selinexor or other XPO1 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Phase 3: Proportion of Participants with Spleen Volume Reduction (SVR) of Greater than or Equal to (>=) 35 Percent (%) (SVR35) at Week 24 Measured by the Magnetic Resonance Imaging (MRI) or Computed Tomography (CT) Scan | At Week 24
Phase 3: Absolute mean change in TSS (Abs-TSS) from baseline to Week 24 as measured by the Myelofibrosis Symptom Assessment Form (MFSAF) v4.0 | At Week 24
Phase 1: Maximum Tolerated Dose (MTD) | Approximately within the first cycle (28 days) of therapy
Phase 1: Recommended Phase 2 Dose (RP2D) | Approximately within the first cycle (28 days) of therapy
Phase 1: Number of Participants With Adverse Events (AEs) by Occurrence, Nature, and Severity | From start of drug administration up to 30 days after last dose of study treatment (approximately 48 months)

SECONDARY OUTCOMES:
Phase 3: Overall survival (OS) | From Baseline up to EoS (approximately 48 months)
Phase 3: Progression-free survival (PFS) | Time from randomization until disease progression or death, whichever occurs first (approximately 48 months)

CONTACTS AND LOCATIONS:
Locations (166):
- United States (36):
  - UAB Division of Hematology/Oncology, Birmingham, Alabama
  - UCLA - Satellite Site, Beverly Hills, California
  - City of Hope, Duarte, California
  - UCLA - Satellite Site, Encino, California
  - City of Hope - Irvine Lennar - Satellite, Irvine, California
  - UCLA, Los Angles, California
  - The Oncology Institute of Hope & Innovation, Pasadena, California
  - USOR - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Smilow Cancer Hospital - New Haven, New Haven, Connecticut
  - Georgetown Lombardi Comprehensive Center, Washington D.C., District of Columbia
  - Norton Cancer Institute - Saint Matthews, Louisville, Kentucky
  - Maryland Oncology Hematology-Satellite, Annapolis, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Maryland Oncology Hematology-Satellite, Brandywine, Maryland
  - Maryland Oncology Hematology, Columbia, Maryland
  - Maryland Oncology Hematology-Satellite, Rockville, Maryland
  - Maryland Oncology Hematology-Satellite, Silver Spring, Maryland
  - The Cancer & Hematology Centers -Satellite Site, Grand Rapids, Michigan
  - The Cancer & Hematology Centers of Muskegon, Norton Shores, Michigan
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Health System, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Institue, Durham, North Carolina
  - USOR - Oncology Hematology Care - Kenwood, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center (OSUCCC) - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - OhioHealth, Columbus, Ohio
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - USOR - Virginia Cancer Specialists - Gainesville Office, Gainesville, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia
  - USOR - Virginia Oncology Associates - Virginia Beach, Virginia Beach, Virginia
  - Fred Hutchinson Cancer Center - SCAA South Lake Union, Seattle, Washington
  - West Virginia University Cancer Institute, Wheeling Hospital, Wheeling, West Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
- Australia (6):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Icon Cancer Centre - Wesley, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - One Clinical Research, Nedlands, Western Australia
- Belgium (5):
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Flemish Brabant
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges, West-Vlaanderen
  - ZNA Stuivenberg - Satelite, Antwerp
  - ZNA Stuivenberg, Antwerp
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment Sveti George - Base 1, Plovdiv
  - University Multiprofile Hospital for Active Treatment Aleksandrovska, Sofia
  - University Multiprofile Hospital for Active Treatment St. Ivan Rilski, Sofia
  - Specialized Hospital for Active Treatment of Hematological Diseases - EAD Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment - Prof. Dr. Stoyan Kirkovich, Stara Zagora
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Lakeridge Health, Oshawa, Ontario
  - Research Institute of the McGill University Health Centre, Montreal, Quebec
- Czechia (3):
  - Vseobecna Fakultni Nemocnice v Praze, Prague, Prague
  - Fakultní Nemocnice Hradec Králové, Hradec Králové
  - Fakultní Nemocnice Olomouc, Olomouc
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus N, Central Jutland
  - Tang Severinsen, Marianne, Aalborg, North Denmark
- France (14):
  - Institut Bergonié, Bordeaux, Aquitaine
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand, Aubergne
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Hôpital Morvan, Brest, Brittany Region
  - Chu De Nîmes - Institut De Cancérologie Du Gard, Nîmes, Gard
  - Hôpital Emile Muller, Mulhouse, Grand Est
  - Hôpital Huriez, Lille, Hauts-de-France
  - Hôpital Bretonneau, Tours, Indre-et-Loire
  - Hôpital l'Archet - CHU Nice, Nice, PACA
  - Centre Hospitalier Universitaire d'Angers, Angers, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Saint-Étienne, Saint-Priest-en-Jarez, Pays de la Loire Region
  - Hôpital Saint-Louis, Paris
  - Hôpital Universitaire Pitié Salpêtrière, Paris, Île-de-France Region
  - Hôpital Cochin, Paris, Île-de-France Region
- Germany (5):
  - Kliniken Ostalb - Stauferklinikum Schwäbisch Gmünd, Mutlangen, Baden-Wurttemberg
  - Marien Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Städtisches Krankenhaus Kiel, Kiel, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia
- Greece (6):
  - Laiko General Hospital of Athens, Athens, Attica
  - General Hospital of Athens "Alexandra", Athens, Attica
  - University General Hospital Attikon, Athens, Attica
  - General Hospital of Thessaloniki George Papanikolaou, Thessaloniki, Central Macedonia
  - University General Hospital of Ioannina, Ioánnina, Thessaly
  - University General Hospital of Larissa, Hematology Department, Larissa, Thessaly
- Hungary (2):
  - Győr-Moson-Sopron Vármegyei Petz Aladár Egyetemi Oktató Kórház, Győr, Győr-Moson-Sopron
  - Semmelweis Egyetem, Budapest
- Israel (9):
  - Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov, Central District
  - The Chaim Sheba Medical Center, Ramat Gan, Central District
  - Rambam Health Care Campus, Haifa, Haifa District
  - Carmel Medical Center, Haifa, Haifa District
  - Hadassah University Hospital - Mount Scopus - Satellite Site, Jerusalem, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem, Jerusalem
  - Emek Medical Center, Afula, Northern District
  - Western Galilee Hospital-Nahariya, Nahariya, Northern District
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (18):
  - Azienda Ospedaliero Universitaria Policlinico Gaspare Rodolico - San Marco - Catania/ Presidio G. Rodolico, Catania, Catania
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST, Meldola, Forli-Cesena
  - IRCCS Ospedale Policlinico San Martino, Genova, Genoa
  - Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico, Milan, Milan
  - Istituto Europeo di Oncologia, Milan, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza and Brianza
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara, Novara
  - IRCCS Centro di Riferimento Oncologico di Basilicata, Rionero in Vulture, Potenza
  - Umberto I - Policlinico di Roma, Roma, Rome
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino, Turin
  - Università Campus Bio-Medico di Roma, Rome, Viterbo
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico Sant Orsola-Malpighi, Bologna
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
  - Centro Ricerche Cliniche di Verona, Verona
- Netherlands (2):
  - Spaarne Gasthuis - Hoofddorp, Hoofddorp, North Holland
  - Universitair Medisch Centrum Groningen, Groningen
- Poland (8):
  - AIDPORT, Skórzewo, Greater Poland Voivodeship
  - Medicover Integrated Clinical Services (MICS) - Centrum Medyczne Toruń, Torun, Kuyavian-Pomeranian Voivodeship
  - Dolnośląskie Centrum Transplantacji Komórkowych z Krajowym Bankiem Dawców Szpiku, Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny Nr 4 w Lublinie, Lublin, Lublin Voivodeship
  - Szpital Specjalistyczny w Brzozowie - Podkarpacki Ośrodek Onkologiczny im. Ks. B. Markiewicza, Brzozów, Podkarpackie Voivodeship
  - Uniwersyteckie Centrum Kliniczne w Gdańsku, Gdansk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice, Katowice, Silesian Voivodeship
  - Specjalistyczny Szpital im. dra Alfreda Sokołowskiego w Wałbrzychu, Wałbrzych, Silesian Voivodeship
- Romania (6):
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca, Cluj
  - Spitalul Filantropia - Craiova, Craiova, Dolj
  - Spitalul Clinic Judetean De Urgenta Târgu Mureș, Târgu Mureş, Mureș County
  - Coltea - Spital Clinic, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Regional De Oncologie Iasi, Iași
- South Korea (8):
  - Pusan National University Hospital, Busan, Gwang'yeogsi
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea - Seoul St. Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (16):
  - Hospital San Pedro de Alcantara, Cáceres, Cáceres
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de Día Quirónsalud Zaragoza, Zaragoza, Zaragoza
  - Institut Català d'Oncologia Badalona, Badalona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Català d'Oncologia Girona (ICO Girona), Girona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Complejo Asistencial Universitario de Salamanca - Hospital Clínico, Salamanca
  - Hospital Clínico Universitario de Valencia, Valencia
- Taiwan (5):
  - China Medical University Hospital, Taichung, Taichung
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District
- United Kingdom (7):
  - Guy's and St Thomas' NHS Foundation Trust, London, England
  - Oxford University Hospitals NHS Foundation Trust, Oxford, England
  - United Lincolnshire Hospitals NHS Trust-Satellite Site, Boston
  - United Lincolnshire Hospitals NHS Trust, Boston
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Imperial College Healthcare NHS Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mascarenhas J, Maher K, Rampal R, Bose P, Podoltsev N, Hong J, Chai Y, Kye S, Method M, Harrison C; SENTRY investigators. Selinexor plus ruxolitinib in JAK inhibitor treatment-naive myelofibrosis: SENTRY Phase 3 study design. Future Oncol. 2025 Mar;21(7):807-813. doi: 10.1080/14796694.2025.2461393. Epub 2025 Feb 6. PMID 39911057